**Title:** Promoting the Application of Tai Chi to Improve the Fatigue in

**Cancer Patients** 

**Protocol ID**:201900504B0

NCT: not yet

## **Study Protocol:**

The purpose of this study is to explore the effectiveness of empirical application of Taichi in improving cancer-related fatigue and other outcome. This research adopts a kind of experimental research design, taking 78 cancer patients hospitalized by traditional Chinese medicine in a teaching area hospital in the Taiwan north as the object, and dividing the cases into two groups. The Taichi group was given routine care and Taijiquan, while the control group was given routine care. After obtaining consent before accepting the case, after the intervention measures started, the pre-test, the first week, the second week, the fourth to the eighth week Follow up and explore the effects of Tai Chi on fatigue, sleep quality, anxiety and depression, heart rate variability, quality of life after intervention.

## **Statistical Analysis Plan (SAP):**

The researcher first checks the integrity of the data, codes the data, and then inputs it into the computer according to the code book. After creating the file, the data is analyzed using IBM SPSS 20.0 software. According to the research purpose and the nature of the variables, the following statistical methods are used to conduct descriptive statistical analysis and inferential statistical analysis. 1. Descriptive statistics include mean, standard deviation, frequency and percentage, and the chi-square test, Fisher's exact test and independent t test are used to detect the homogeneity of the basic attributes and clinical disease characteristics of the two groups. sex. 2. Inferential statistics used Repeat Measure ANOVA to analyze the effect of Tai Chi health intervention time on fatigue, sleep quality, quality of life and heart rate variability. In this study, P <0.05 was considered as a statistically significant difference.